CLINICAL TRIAL: NCT03762655
Title: Randomized, Controlled, Single-blind Study of Probable Benefit of the Neuro-Spinal Scaffold™ for Safety and Neurologic Recovery in Subjects With Complete Thoracic AIS A Spinal Cord Injury as Compared to Standard of Care
Brief Title: Study of Probable Benefit of the Neuro-Spinal Scaffold™ in Subjects With Complete Thoracic AIS A Spinal Cord Injury as Compared to Standard of Care
Acronym: INSPIRE 2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary Endpoint not met
Sponsor: InVivo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: InVivo-100-105
Record Dates: First submitted 2018-11-29; First posted 2018-12-04 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2022-06

CONDITIONS: Injury, Spinal Cord
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a blinded manner to one of two study arms, the Treatment or "Scaffold" Arm and the Standard of Care or "Comparator" Arm. Subjects in the Scaffold Arm will have the Scaffold implantation immediately following standard of care open spine surgery. Subjects in the Comparator Arm will have standard of care open spine surgery and will not receive the Scaffold.
Who Masked: Participant
Masking Description: Subjects will be randomized in a blinded manner to one of two study arms, the Treatment or "Scaffold" Arm and the Standard of Care or "Comparator" Arm. Subjects in the Scaffold Arm will have the Scaffold implantation immediately following standard of care open spine surgery. Subjects in the Comparator Arm will have standard of care open spine surgery and will not receive the Scaffold. The subjects will be blinded to their study arm for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Neuro-Spinal Scaffold Arm (Experimental): Subjects in the Scaffold Arm will have the Scaffold implantation immediately following standard of care open spine surgery.
  Interventions: Device: Neuro-Spinal Scaffold
- Comparator Arm (No Intervention): Subjects in the Comparator Arm will have standard of care open spine surgery and will not receive the Scaffold.

INTERVENTIONS:
Device: Neuro-Spinal Scaffold — The investigational product ("Neuro-Spinal ScaffoldTM" or "Scaffold") is a porous bioresorbable polymer scaffold comprised of a synthetic biomaterial, poly(lactic-co-glycolic acid)-b-poly(L-lysine) (PLGA-PLL). The Scaffold is cylindrical in shape (3 mm diameter) and is available is three lengths (6 mm, 8 mm, 10 mm) for optimal fit in the intraspinal lesion cavity.
  Based upon pre-clinical testing, the Scaffold is expected to be resorbed from the site of implant within 4 to 8 weeks.
  Arms: Neuro-Spinal Scaffold Arm

SUMMARY:
This is a randomized, controlled, single-blind, multicenter, two Arm (Treatment or "Scaffold" Arm; Standard of Care or "Comparator" Arm) of a Neuro-Spinal Scaffold to evaluate whether the Scaffold is safe and demonstrates probable benefit for the treatment of complete T2-T12 spinal cord injury as compared to standard of care open spine surgery.

DETAILED DESCRIPTION:
This is a randomized, controlled, single blind, two-arm, multicenter Humanitarian Device Exemption (HDE) study to evaluate the safety and probable benefit of the poly(lactic-co-glycolic acid)-b-poly(L-lysine) Scaffold ("Scaffold") in subjects with thoracic AIS A traumatic spinal cord injury at neurological level of injury of T2-T12 as compared to standard of care open spine surgery. Subjects will be randomized in a blinded manner to one of two study arms, the Treatment or "Scaffold" Arm and the Standard of Care or "Comparator" Arm. Subjects in the Scaffold Arm will have the Scaffold implantation immediately following standard of care open spine surgery. Subjects in the Comparator Arm will have standard of care open spine surgery and will not receive the Scaffold. The subjects will be blinded to their study arm for the duration of the study.

Primary Objective: To evaluate whether the Scaffold is safe and demonstrates probable benefit for the treatment of complete T2-T12 spinal cord injury as compared to standard of care open spine surgery.

Regulatory Objective: To enhance the clinical evidence for the Scaffold in the treatment of complete thoracic spinal cord injuries.

Intended Use: The Scaffold is intended for use in patients age 16-70 years diagnosed with a T2-T12 neurological level of injury functionally complete (AIS A) spinal cord injury for whom open spine surgery, (e.g., laminectomy, spine stabilization) which allows access to the dura of the injured spinal cord, is recommended as an option. The Scaffold is intended to be implanted in a cavity at the epicenter of the spinal cord contusion during open spine surgery. The Scaffold is intended for use in recent (≤7 days) spinal cord injuries that do not involve penetrating injury to the cord or complete severing of the cord.

ELIGIBILITY:
Inclusion Criteria:

1. AIS A classification of traumatic spinal cord injury at T2 - T12 neurological level of injury confirmed by a qualified medical professional
2. Recent injury (must have open spine surgery within 7 days from injury)
3. Injury Severity Score (ISS) ≤ 45 at the time of screening
4. Glasgow Coma Scale, GCS ≥ 14 (GCS ≥ 10 for intubated subjects) at the time of the screening and GCS = 15 (GCS ≥ 10 for intubated subjects) within two hours prior to spine surgery
5. Non-penetrating SCI (contusion injury) that is no less than approximately 4 mm in diameter by MRI
6. Requires open spine surgery allowing access to the injured spinal cord (subjects requiring either posterior surgical approach or posterior plus anterior approach will be eligible)
7. Informed consent obtained
8. 16-70 years of age, inclusive
9. Eight-hour period of hemodynamically stability (>90 mmHg systolic blood pressure) prior to open spine surgery

Exclusion Criteria:

1. Terminally ill subjects not likely to be able to participate in follow-up
2. Incomplete spinal cord injury (AIS B, C, D, and E injuries)
3. Subjects with more than one discrete spinal cord injury
4. No discrete cavity in the contused spinal cord in which a Scaffold can be placed
5. Evidence of clear and significant Somatosensory Evoked Potentials (SSEP) transmission through the injury site (based on the judgment of the Investigator)
6. Subjects with clinically significant pre-existing neurological comorbidities that are unrelated to the contusion being treated (e.g. MS, ALS, significant prior peripheral nerve dysfunction, residual problems related to previous spine-related neurological pathologies) will be excluded only if it is felt that these preexisting morbidities will increase risk, affect safety monitoring, or confound study results
7. Spinal cord injury associated with significant traumatic brain injury or coma that, in the opinion of the Investigator, would preclude adequate assessment of spinal cord function, brain injury that could be associated on its own with sensory or motor deficits, or subjects with any other reason that results in an unreliable ISNCSCI exam
8. Subjects with clinically significant pre-existing respiratory disease not related to the contusion being treated (e.g., COPD)
9. Subjects requiring long-term ongoing mechanical ventilation
10. Subjects with documented immune deficiency disorders, including a known diagnosis of HIV infection/AIDS
11. Recent (according to DSM IV or DSM V criteria) history of abuse of narcotics or other significant substance abuse
12. Significant injury complications where, in the view of the Investigator, participation in the study could further complicate subject care, limit study follow-up, or confound interpretation of safety or efficacy data.
13. A female who is:

    * Pregnant, or planning to become pregnant within the next 12-months; or
    * Breastfeeding; or
    * A woman of child-bearing potential (defined as post menarche and biologically capable of becoming pregnant [i.e., not surgically sterile]) who is engaged in active heterosexual relations and is not willing to use a barrier or hormonal form of birth control for 12-months following open spine surgery (e.g., oral, injected, or implanted contraceptives)
14. A male who is engaged in active heterosexual relations and is not willing to use birth control for 3-months following open spine surgery including sperm donation or banking
15. Current or impending incarceration
16. Complete spinal cord transection as determined by screening MRI
17. Subjects with spinal cord injuries directly due to gunshot, knife, or other penetrating wounds.
18. Known hypersensitivity to PLGA or PLL (e.g., hypersensitivity to absorbable sutures containing PLGA)
19. History of severe mental illness (according to DSM IV or V)
20. Evidence of pre-trauma active local or systemic infection
21. Participation in another interventional clinical trial for six months after open spine surgery
22. BMI over 39
23. Having a medical condition (e.g., cardiovascular disease, life threatening injuries), or receiving medical treatment, or having any other reason that, in the judgment of the Investigator, precludes successful participation and follow-up for at least six months or confounds collection or interpretation of study safety, feasibility, or efficacy data
24. Subjects receiving tetracyclines, such as minocycline (subjects must discontinue tetracyclines to be enrolled in the study; tetracyclines can be resumed after 6 months post-open spine surgery

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in AIS grade of one or more levels | 6 months post-implant
  The proportion of subjects with an improvement of at least one AIS grade will be presented for each study arm.
  The International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) examinations determine the ASIA Impairment Scale (AIS) grade.

SECONDARY OUTCOMES:
Change in Neurological Level of Injury (NLI) | 3-months, 6-months, 12-months, 24-months post-open spine surgery
  The ISNCSCI examinations determine the the Neurological Level of Injury (NLI). The NLI refers to the most caudal segment of the spinal cord with normal sensory and antigravity motor function on both sides of the body, provided that there is normal (intact) sensory and motor function rostrally.
  NLI will be summarized for each study arm at visits (pre-surgery, 3-months, 6-months, 12-months, 24-months). Observed values and change from the baseline will be presented for each study arm.The ISNCSCI exam performed within 8 hours prior to surgery (pre-surgery ISNCSCI) will be used as the baseline.
Change in motor scores | 3-months, 6-months, 12-months, 24-months post-open spine surgery
  A numerical summary score of motor function in each extremity determined by the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) examination. This score can reflect the degree of neurological impairment associated with the SCI, with lower score indicating greater impairment. Score ranges from 0-25 for each extremity, with maximum scores of 50 for the upper limbs and 50 for the lower limbs.
  Motor scores will be summarized for each study arm at visits (pre-surgery, 3-months, 6-months, 12-months, 24-months). Observed values and change from the baseline will be presented for each study arm.The ISNCSCI exam performed within 8 hours prior to surgery (pre-surgery ISNCSCI) will be used as the baseline.
Change in sensory scores | 3-months, 6-months, 12-months, 24-months post-open spine surgery
  A numerical summary score of sensory function in each determined by the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) examination. This score can reflect the degree of neurological impairment associated with the SCI, with lower score indicating greater impairment. Score ranges from 0-56 points each for light touch and pin prick (sharp/dull discrimination) modalities, with a maximum total score of 112 points per side of the body.
  Observed values and change from the baseline will be presented for each study arm.The ISNCSCI exam performed within 8 hours prior to surgery (pre-surgery ISNCSCI) will be used as the baseline.
Changes in bladder, bowel, and sexual function | 6-months, 12-months and 24-months, post-open spine surgery
  Bladder, bowel and sexual function will be assessed using the Lower Urinary Tract, Bowel and Sexual Function System/Organ section of the ASIA Autonomic Standards Assessment Form. The Autonomic Standards Assessment Form has three questions in each category (Lower Urinary Tract or bladder, Bowel, Sexual Function) and each question is scored on a scale from 0 (complete loss of control) - 2 (normal function). Observed values and change from baseline will be presented for each study arm. The hospital discharge visit will be used as the baseline visit.
Changes in spinal cord dimension | 72-hours, 3-months, 6-months, 12-months, and 24-months post-open spine surgery
  Spinal cord dimensions (above, at, and below level of injury) will be assessed by an independent board-certified neuroradiologist central reader. Observed values and change from baseline will be presented for each study arm. The Screening MRI will be used as the baseline.
Changes in spinal cord lesion size | 72-hours, 3-months, 6-months, 12-months, and 24-months post-open spine surgery
  Lesion size (in mm) will be assessed by an independent board-certified neuroradiologist central reader. Observed values and change from baseline will be presented for each study arm. The Screening MRI will be used as the baseline.
Changes in spinal cord lesion location | 72-hours, 3-months, 6-months, 12-months, and 24-months post-open spine surgery
  Lesion Location will be assessed by an independent board-certified neuroradiologist central reader. Observed values and change from baseline will be presented for each study arm. The Screening MRI will be used as the baseline.
Changes in spinal cord anatomy-Presence of cyst | 72-hours, 3-months, 6-months, 12-months, and 24-months post-open spine surgery
  Cyst presence or absence will be assessed by an independent board-certified neuroradiologist central reader. Observed values and change from baseline will be presented for each study arm. The Screening MRI will be used as the baseline.
Changes in cyst size, if present | 72-hours, 3-months, 6-months, 12-months, and 24-months post-open spine surgery
  Cyst size, if present, will be assessed by an independent board-certified neuroradiologist central reader. Observed values and change from baseline will be presented for each study arm. The Screening MRI will be used as the baseline.
Changes in cyst location, if present | 72-hours, 3-months, 6-months, 12-months, and 24-months post-open spine surgery
  Cyst location, if present, will be assessed by an independent board-certified neuroradiologist central reader. Observed values and change from baseline will be presented for each study arm. The Screening MRI will be used as the baseline.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - UC Davis Medical Center, Sacramento, California
  - University of California San Diego, San Diego, California
  - University of Colorado Memorial Hospital Central, Colorado Springs, Colorado
  - University of South Florida Health Neurosurgery, Tampa, Florida
  - University of Iowa, Iowa City, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Rutgers Center for Spine Surgery, Newark, New Jersey
  - Elmhurst Hospital Center, Elmhurst, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Vidant Medical Center, Greenville, North Carolina
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center-Presbyterian, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Texas Health San Antonio, San Antonio, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Harrop JS, Kim KD, Okonkwo DO, Goldstein IM, Lee KS, Toselli RM. Acute Implantation of a Bioresorbable Polymer Scaffold in Patients With Complete Thoracic Spinal Cord Injury: A Randomized Controlled Trial (INSPIRE 2.0). Neurosurgery. 2025 Apr 1;96(4):751-762. doi: 10.1227/neu.0000000000003180. Epub 2024 Oct 8. PMID 39471088